CLINICAL TRIAL: NCT01689181
Title: L'apathie Dans La Schizophrénie: Étude Neuropsychologique Et Anatomique
Brief Title: Apathy in Schizophrenia
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C11-39; 2011-A01610-41 (Registry Identifier: IDRCB)
Record Dates: First submitted 2012-09-07; First posted 2012-09-21 (Estimated); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Schizophrenia; Apathy
MeSH Terms: conditions — Schizophrenia; Lethargy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- chronic schizophrenic patients
- healthy volunteers

SUMMARY:
Apathy, defined as a quantitative reduction of voluntary, goal-directed behaviours (GDB), is a core component of negative symptoms. It has been suggested that the physiopathology of apathy is not a single entity but may be multiple, depending on which specific process or macrofunction is disrupted during completion of GDB. In line with this notion, Levy and Dubois proposed dividing apathic syndromes into three subtypes of disrupted processing: 'a-motivation', 'cognitive inertia', and 'uncoupling'. In schizophrenia, apathy has been associated with executive dysfunction, functional impairment and poor outcome. However, the neurobiological underpinnings of apathy in schizophrenia are poorly understood.

Primary objective: confirm that chronic schizophrenic patients are apathic compared to healthy volunteers

Secondary objectives:

* investigate if apathy is related to a particular aspect of the disease (i.e. negative, positive symptomatology and/or deficit form)
* investigate if apathy correlates with executive dysfunction
* investigate if apathy is associated with a specific mechanism using an experimental task specially designed to investigate the different mechanism (i.e. 'a-motivation', 'cognitive inertia', and 'uncoupling')
* investigate if there is a volumetric abnormality affecting the executive system in apathic schizophrenic patients
* link these eventual volumetric abnormalities to prefrontal cortex-basal ganglia circuits according to a specific subtype of apathy in the apathic schizophrenic group

ELIGIBILITY:
Inclusion Criteria (healthy volunteers):

* Male or Female aged 20 to 55 years old included
* Under French public assurance system

Exclusion Criteria (healthy volunteers):

* Personal history of neurological disorders
* Personal history of head injury
* Alcohol or substance abuse
* Under psychotropic drug
* Contraindication for MRI

Inclusion Criteria (schizophrenic patients):

* Male or Female aged 20 to 55 years old included
* Under French public assurance system
* diagnosis of schizophrenia according to the DSM-IV R criteria
* Duration of illness > 5 years
* clinical stability during the past 2 months (defined as no treatment modification or hospitalisation 2 months prior evaluation)

Exclusion Criteria (schizophrenic patients):

* Schizo-affective disorder
* Personal history of neurological disorders
* Personal history of head injury
* Alcohol or substance abuse
* Contraindication for MRI

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: schizophrenic patients:
  * outpatients of the Corentin Celton psychiatric service
  * inpatients of the Corentin Celton Day Hospital Unit
  healthy volunteers: community
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2013-06-05 (Actual); Study Completion 2013-06-05 (Actual)

PRIMARY OUTCOMES:
apathy as measured by Starkstein's Apathy Evaluation Scale | baseline

SECONDARY OUTCOMES:
neuropsychological performance | baseline
  * Global mental efficience: Mill Hill B and Raven's progressive matrices 38
  * Executive functioning:Modified Card Sorting Test, Trail Making A and B, Stroop Test, Verbal Fluences, Frontal Assessment Battery (FAB, Dubois et al., 2000)
  * Social and Emotional Cognition: SEA (Social and Emotional Evaluation (SEA, Funkiewiez et al., 2012)
  * Working memory (Grober and Buschke - 16 items, digit span)
  * Instrumental functions: Rey Osterrieth Complex figure)
clinical assessment (for patients only) | baseline
  scores on evaluation scales (PANSS, SAPS, SANS, CDS, SDS)
volumetric brain abnormalities | baseline
  voxel based morphometry

CONTACTS AND LOCATIONS:
Overall Officials: Richard Levy, MD, Principal Investigator — INSERM MEDU 945, Centre de Recherche-Institut du Cerveau et de la Moelle (CR-ICM), Hôpital de la Pitié Salpétrière, 75013 Paris
Locations (1):
- INSERM MEDU 945, Centre de Recherche-Institut du Cerveau et de la Moelle (CR-ICM), Hôpital de la Pitié Salpétrière, Paris, France